CLINICAL TRIAL: NCT06776510
Title: A Prospective, One-arm and Open Clinical Study to Assess Safety and Efficacy of Nicotinamide Adenine Dinucleotide in the Treatment of Primary Immune Thrombocytopenia
Brief Title: A Clinical Study of NAD in the Treatment of Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024089
Record Dates: First submitted 2025-01-07; First posted 2025-01-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Nicotinamide Mononucleotide; NAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: (Experimental): nicotinamide adenine dinucleotide/nicotinamide mononucleotide
  Interventions: Drug: nicotinamide adenine dinucleotid/nicotinamide mononucleotide

INTERVENTIONS:
Drug: nicotinamide adenine dinucleotid/nicotinamide mononucleotide — Drug: intravenous nicotinamide adenine dinucleotide (Coenzyme I for Injection) administration This study adopts a prospective, single arm, open design method. Twenty subjects were enrolled in the study and were treated with nicotinamide adenine dinucleotide (100mg/d) for 1 week.
  Drug: oral nicotinamide mononucleotide administration This study adopts a prospective, single arm, open design method. Twenty subjects were enrolled in the study and were treated with nicotinamide mononucleotide 450mg BID for 2 weeks.
  The first stage is the main research stage (d0-w2), which is the core treatment period. The aim is to observe the safety and efficacy during treatment.
  The second stage (w2-w8) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy after treatment.
  Other Names: Coenzyme I for Injection（NAD+）/NMN

SUMMARY:
To evaluate the safety and efficacy of nicotinamide adenine dinucleotide in the treatment of immune thrombocytopenia in patients who have not responded adequately or relapsed after first-line treatment and at least one second-line therapy including Anti-CD20 Antibody and/or TPO-RA.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. However, targeting LLPC becomes a new strategy to treat autoimmune diseases.

CM313, a kind of anti-CD38 antibody, is a new type of monoclonal antibody targeting CD38. It targets plasma cells and has carried out some clinical studies in multiple myeloma, with good therapeutic effects. We treated patients with refractory/relapsed ITP using CM313 and achieved good therapeutic outcomes, which may provide a new strategy for treating ITP. Current research shows that CD38, as a metabolic enzyme, can hydrolyze nicotinamide adenine dinucleotide (NAD+), leading to a decrease in intracellular NAD+. Additionally, during aging and inflammation, CD38 is highly expressed on macrophages, and the downregulation of NAD+ levels. Based on the current mechanistic studies of CD38 monoclonal antibody treatment for ITP, we found that macrophages in ITP patients exhibit a shift towards M1 polarization. We hypothesize that CD38 antibodies may reduce platelet destruction by macrophages by upregulating NAD+ levels, which in turn inhibits M1 polarization. Therefore, increasing NAD+ levels may have therapeutic potential for ITP. Since nicotinamide adenine dinucleotide (NAD+) has been used in clinical practice as an adjunctive treatment for leukopenia, coronary artery disease as well as myocarditis, and nicotinamide mononucleotide (NMN) has been explored in clinical trials, we will further investigate the therapeutic efficacy and safety of these compounds in ITP patients.

Therefore, the investigators designed this clinical trial to evaluate the safety and efficacy of Nicotinamide Adenine Dinucleotide (Coenzyme I for Injection, NAD+) and nicotinamide mononucleotide (NMN) in the treatment of primary immune thrombocytopenia in patients who are steroid-refractory or steroid-dependent, and fail to respond to at least one previous second-line therapy, including rituximab and/ or TPO agonist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female;
* Conform to the diagnostic criteria of immune Thrombocytopenia (ITP) ≥3 months;
* Failure to achieve response or relapse after corticosteroid therapy, and failure to achieve response or relapse after previous second-line treatments such as TPO/TPORAs therapy, or are unable to afford the cost of the treatment;
* The platelet count of <30 X 10^9/L measured within 2 days prior to inclusion (During the screening visit and/or before receiving the study drug, platelet counts must be less than 30×10^9/L on at least two consecutive occasions, with a minimum interval of 1 day between the two tests.);
* ECOG physical state score ≤ 2 points;
* Subjects on stable dose maintenance therapy are allowed to be included (concomitant medications may include corticosteroids (≤0.5 mg/kg of prednisone or equivalent steroids) or TPO receptor agonists, etc.), but at the time of enrollment, only one concomitant medication with a stable dose is permitted. The concomitant medication must have been on a stable dose for at least 4 weeks prior to the first dose of the study drug;
* For female patients of childbearing potential, a negative pregnancy test result is required. Both female patients of childbearing potential and male patients must use highly effective contraception during the study and for 4 months/6 months after discontinuing treatment;
* Signed and dated written informed consent

Exclusion Criteria:

* Those who are allergic to Nicotinamide adenine dinucleotide or excipients, or who have previously received CD38 monoclonal antibody treatment with no efficacy.
* Those with autoimmune hemolytic anemia, or various types of secondary and genetic thrombocytopenia, such as leukemia, lymphoma, multiple myeloma, aplastic anemia, myelodysplastic syndrome, Evans syndrome, common variable immunodeficiency, systemic lupus erythematosus, cirrhosis, antiphospholipid antibody syndrome, pseudo-thrombocytopenia, drug-induced thrombocytopenia (e.g., quinine, heparin, antimicrobial drugs, anticonvulsants, etc.).
* A history of any thrombosis or embolism events within 12 months prior to the first dose, or the presence of extensive and severe bleeding, such as hemoptysis, upper gastrointestinal bleeding, intracranial hemorrhage, sepsis, or other irregular bleeding.
* Participation in any other clinical trial involving investigational drugs (including vaccine studies) or exposure to other investigational drugs within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose.
* Use of anticoagulants or any drugs with antiplatelet effects (e.g., aspirin) within 2 weeks prior to the first dose.
* Receiving emergency treatment for ITP within 2 weeks prior to the first dose (e.g., methylprednisolone, platelet transfusion, intravenous immunoglobulin, or TPO receptor agonist treatment).
* Receiving azathioprine, danazol, cyclosporine A, tacrolimus, sirolimus, or similar drugs within 4 weeks prior to the first dose; receiving CD20 monoclonal antibodies such as rituximab, cyclophosphamide, vincristine, or similar drugs within 3 months prior to the first dose.
* Splenectomy within 6 months prior to the first dose.
* Receiving a live vaccine within 4 weeks prior to the first dose, or planning to receive any live vaccine during the study period.
* A history of undergoing allogeneic stem cell transplantation or organ transplantation.
* A history of clinically significant diseases that, in the investigator's opinion, may pose a risk to the subject's safety or affect the assessment of safety or efficacy during the study if the disease/condition worsens.
* Subjects who have had malignant tumors within the past 5 years prior to screening (excluding completely cured carcinoma in situ of the cervix and non-metastatic squamous cell carcinoma or basal cell carcinoma of the skin).
* Exhibiting clinically significant laboratory abnormalities at screening: a) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ the upper limit of normal (ULN); b) Total bilirubin ≥ 1.2 times ULN. ;c) Creatinine or blood urea nitrogen (BUN) ≥ ULN.
* Positive for HIV antibodies or syphilis antibodies.
* Positive for hepatitis B surface antigen (HBsAg) at screening, or positive for hepatitis B core antibody with a positive HBV-DNA result by polymerase chain reaction (PCR) testing, or positive for hepatitis C virus (HCV) antibodies.
* Women who are pregnant or breastfeeding, or planning to become pregnant or breastfeed during the study; and men whose partners are planning to become pregnant during the study.
* Subjects with mental disorders who are unable to provide informed consent or participate in the trial and follow-up properly.
* Subjects with unresolved toxicity symptoms caused by prior treatments before participating in the trial.
* Any other conditions deemed unsuitable for participation in this study as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of overall efficacy response after nicotinamide adenine dinucleotide/NMN treatment within 2 weeks | [Time Frame: 2 weeks]
  Proportion of subjects with a platelet count ≥ 50 × 10^9/L (two consecutive measurements at least 1 day apart) within 2 weeks after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
incidence of treatment-emergent Adverse Events and TRAE | [Time Frame: 8 weeks]
  Incidence, severity, and relationship of treatment emergent adverse events after nicotinamide adenine dinucleotide/NMN treatment

SECONDARY OUTCOMES:
Evaluation of the efficacy at each visit period | [Time Frame: 8 weeks]
  Proportion of subjects with a platelet count ≥ 50 × 10^9/L at week 1, week 2, week 3, week 4, week 6，week 8 in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Duration from treatment initiation to platelet count ≥30×10^9/L (at least two times of baseline platelet count) and ≥50×10^9/L | [Time Frame: 8 weeks]
  Duration from treatment initiation to platelet count ≥30×10^9/L (at least two times of baseline platelet count) and ≥50×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
Platelet count at each visit time point | [Time Frame: 8 weeks]
  Platelet count values at each visit time point including day0, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8.
Emergency treatment | [Time Frame: 8 weeks]
  The proportion of subjects who received emergency treatment within 2 weeks and during the entire study period.
Cumulative weeks of platelet ≥30×10^9/L (at least two times of baseline platelet count) and platelet ≥50×10^9/L | [Time Frame: 8 weeks]
  Cumulative weeks of platelet ≥30×10^9/L (at least two times of baseline platelet count) and platelet ≥50×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
The change in bleeding score before treatment and 2 weeks after treatment assessed using the world health organization (WHO) bleeding scale | [Time Frame: 2 weeks]
  The change in bleeding score before treatment and 2 weeks after treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Evaluation of the efficacy during the first 4 weeks | 4 weeks
  Proportion of subjects achieving platelet counts ≥ 50×10^9/L at least once in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the first 4 weeks
The response rate within 4 weeks | 4 weeks
  Proportion of subjects whose platelet counts ≥ 30×10^9/L and at least two times of baseline platelet count in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids within 4 weeks（two consecutive measurements at least 7 days apart）.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI